CLINICAL TRIAL: NCT01708018
Title: Pilot Study: Effects of Relaxing Hydrotherapy WATSU in Third Trimester of Pregnancy, an Explorative Cohort-Study
Brief Title: Effects of Relaxing Hydrotherapy in Third Trimester of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: BFH Berner Fachhochschule für Gesundheit (Unknown); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 058/12; Studytyp A, Nr. 2211; SAP-Fall-Nr.: 3991344; SAP-Patient: 11095660
Record Dates: First submitted 2012-10-08; First posted 2012-10-16 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy; Breech Presentation; Low Back Pain; Stress, Psychological
Keywords: Pregnancy; Stress, Psychological; Low Back Pain; Breech Presentation; Relaxation; Hydrotherapy; Acupressure; WATSU
MeSH Terms: conditions — Breech Presentation; Low Back Pain; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Prior and post intervention period (on days 1 and 4) and final control (day 8): ultrasound examination of position of the fetus and amount of amniotic fluid. On these days plus weekly (until birth) questionnaires (QoL: SF-36, EQ-5D-5L, stress: PSS, psychological wellbeing: MDBF, current stress and pain: VAS). Survey concerning birth.
- Intervention group (Experimental): Prior and post intervention (days 1 and 4) and final control (day 8): ultrasound examination of position of the fetus and amount of amniotic fluid. On these days plus weekly (until birth) questionnaires (QoL: SF-36, EQ-5D-5L, stress: PSS, psychological wellbeing: MDBF, current stress and pain: VAS). After the second intervention(day 4): qualitative questionnaire for intervention-group only. Survey concerning birth.
  Interventions: Procedure: WATSU

INTERVENTIONS:
Procedure: WATSU — WATSU (WaterShiatsu) is a gentle form of hydrotherapy that was established in the 1980s. The standardized 60min-intervention applied in this trial is called WATSU-Transition-Flow (Dull, 1997) and is adapted for the third trimester. The mother's abdomen is not being touched during the treatment.
  The treatment takes place in a one-to-one hands-on-setting in the warm- water-therapy-pool (35°C, 95°F) of the University Hospital in Bern and consists of acupressure massage according to the Japanese massage-technique Shiatsu, in an attempt to harmonize the mother's "energy-flow" in the so called "meridians" (energy-channels) of Traditional Chinese Medicine. These "meridians" are also sought to be influenced by slow passive stretches of the mother's extremities. In addition, mobilization of her spine is being enhanced by gravity-free movements.
  During the study, each participant in the intervention group will be treated twice with WATSU (60min treatment at day 1 and 4).
  Arms: Intervention group

SUMMARY:
This study will be the first scientific approach to investigate physical and psychological effects of the passive hydrotherapy-method WATSU (WaterShiatsu) on women and their unborn children at the third trimester of pregnancy. Potential therapeutic benefits of the method shall be evaluated.

It is being hypothesized that WATSU is related to measurable changes in everyday stress perception, psychological wellbeing, quality of life, pregnancy-related low back pain, tonus of the uterus, amount of amniotic fluid, spontaneous course of breech presentations, prospects of external cephalic versions.

Participants in the intervention-group will be treated twice with WATSU (60 minutes per treatment, standardized sequence) in the >36th week of pregnancy. There will not be any sham-intervention in the control-group. Both groups will be examined by ultrasound (prior and after the treatments plus on day 8 of the trial) and answer questionnaires (prior and after the treatments plus once a week until birth).

DETAILED DESCRIPTION:
Background

Within the last 20 years, evidence supporting harmlessness and benefits of hydrotherapy during pregnancy accumulated. Water gymnastics were observed to have pain-relieving effects, as was birth in water.

WATSU is an acronym, based on the terms Water and Shiatsu. It is a relaxing form of hydrotherapy which is performed in 35° C (95° F). Practitioners claim WATSU to lower muscular tonus as well as stress and to relief pain. Clinically relevant regulation of muscular tonus in spastic hemiparetic patients due to WATSU was observed by Chon; significant reduction of pain in patients suffering fibromyalgia by Faull.

In respect of pregnancy, WATSU is narrated - yet not scientifically evaluated - to reduce pregnancy-related low back pain, to relax hypertonic muscles including those of the uterus, to improve the overall sense of wellbeing and deepen the relationship of the mother to her unborn child. In addition, spontaneous cephalic versions of children in breech presentations within 1 to 4 days and nights following WATSU-treatments are being claimed.

According to Pennick & Young, two of three pregnant women are suffering pregnancy-related low back pain. Since this population is recommended to refrain from analgesic medications, potentially helpful interventions ought to be identified.

The described effects of WATSU on muscle tone might be of interest in case of breech presentations. Tension of the uterus has major influence on the success of attempts of external cephalic version. Although breech presentation occurs in 3-4% of pregnancies only, this complication is a threat to the mothers as well as the infants life. External cephalic version to correct the child's position is being suggested although associated with risks for mother and child. Breech presentations are the most frequent medical indication for cesarean sections.

The impacts of stress on unborn children are being investigated, long-term effects are being speculated.

Objective

In contrast to active hydrotherapy, passive hydrotherapy was not yet subject of investigation concerning its effects during pregnancy. The goals of this pilot-study are:

* To evaluate the effects of passive hydrotherapy WATSU in the third trimester of pregnancy by the means of a scientific prospective approach and to ascertain, whether the reported effects can be observed under such conditions
* To evaluate the therapeutic potential of WATSU
* To evaluate the usefulness, feasibility and framework requirements of further RCT addressing this issue
* To evaluate, whether or not - which of, respectively - the chosen parameter are suitable for further investigations (RCT)
* To evaluate potential for improvement in study design and management.

Methods

Design: pilot-study, explorative comparison of two cohorts. Criterion for pseudorandomisation: immersion contraindicated (e.g. due to perforation of the eardrum). Recruitment from July to December 2012; expected participants: 45.

Parameter: ultrasound examination of position of the fetus and amount of amniotic fluid; qualitative and quantitative questionnaires, birth outcome (vaginal, cesarean, complications, breech presentation).

Statistics: SPSS; significance at p<.05, Intention to Treat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* singleton pregnancy
* without pathological findings
* at week of gestation >36+0
* fluent German
* Pregnancy related low back pain
* breech presentation
* written informed consent

Exclusion Criteria

* Neurological deficits resulting from low back pain
* already ongoing WATSU-treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in psychological stress | Day 8

SECONDARY OUTCOMES:
Low back pain | Days 1, 4, 8, and weekly until birth
Breech presentation | Days 1, 4, 8, and weekly until birth
Quality of Life | Days 1, 4, 8, and weekly until birth
Amount of amniotic fluid | Days 1, 4, 8
Qualitative questionnaire | Day 4
Birth (vaginal, cesarean, complications, breech) | after birth
Psychological wellbeing | Days 1, 4, 8 and weekly until birth

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Prof. Dr. med., Study Chair — Department of Obstetrics and Gynecology, University Hospital Bern; Luigi Raio, PD Dr. med., Study Director — Department of Obstetrics and Gynecology, University Hospital Bern; Agnes M Schitter, MSc PT, Study Director — BFH Bern University of Applied Sciences
Locations (1):
- Department of Obstetrics and Gynecology, University Hospital, Inselspital, Effingerstrasse 102, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Schitter AM, Nedeljkovic M, Baur H, Fleckenstein J, Raio L. Effects of Passive Hydrotherapy WATSU (WaterShiatsu) in the Third Trimester of Pregnancy: Results of a Controlled Pilot Study. Evid Based Complement Alternat Med. 2015;2015:437650. doi: 10.1155/2015/437650. Epub 2015 Mar 1. PMID 25815033
- See also: Link to trial on the official website of the association of practitioners of WATSU in Switzerland — http://www.iaka.ch/studien